CLINICAL TRIAL: NCT04744831
Title: A Phase 2, Multicenter, Randomized, Study of Trastuzumab Deruxtecan in Participants With HER2-overexpressing Locally Advanced, Unresectable or Metastatic Colorectal Cancer (DESTINY-CRC02)
Brief Title: Trastuzumab Deruxtecan in Participants With HER2-overexpressing Advanced or Metastatic Colorectal Cancer
Acronym: DESTINY-CRC02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS8201-A-U207; 2020-004782-39 (EudraCT Number)
Record Dates: First submitted 2021-01-19; First posted 2021-02-09 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Advanced Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; HER2 Overexpressing Colorectal Cancer; BRAF Wild-Type Status; DS-8201a; Trastuzumab deruxtecan; Advanced Colorectal Cancer; T-DXd
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T-DXd 5.4 mg/kg Q3W (Experimental): Participants will be randomized to receive intravenous T-DXd administered at a dose of 5.4 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: DS-8201a 5.4 mg/kg Q3W
- T-DXd 6.4 mg/kg Q3W (Experimental): Participants will be randomized to receive intravenous T-DXd administered at a dose of 6.4 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: DS-8201a 6.4 mg/kg Q3W

INTERVENTIONS:
Drug: DS-8201a 5.4 mg/kg Q3W — DS-8201a for injection will be administered intravenously (IV) at a dose of 5.4 mg/kg every 3 weeks (Q3W)
  Other Names: T-DXd
  Arms: T-DXd 5.4 mg/kg Q3W
Drug: DS-8201a 6.4 mg/kg Q3W — DS-8201a for injection will be administered intravenously (IV) at a dose of 6.4 mg/kg every 3 weeks (Q3W)
  Other Names: T-DXd
  Arms: T-DXd 6.4 mg/kg Q3W

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of Trastuzumab deruxtecan (T-DXd) in participants with human epidermal growth factor 2 (HER2)-overexpressing locally advanced, unresectable, or metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
This 2-stage study will evaluate participants with locally advanced, unresectable, or metastatic HER2-overexpressing colorectal cancer (CRC) (immunohistochemistry [IHC] 3+ or IHC 2+/ in situ hybridization [ISH]+) of v-raf murine sarcoma viral oncogene homologue B1 (BRAF) wild-type and either rat sarcoma viral oncogenes homologue (RAS) wild-type or mutant tumor type, previously treated with standard therapy. In the first stage, participants will be randomized 1:1 with 2 doses of T-DXd. After Stage 1 enrollment is complete, all further eligible participants will be registered to T-DXd administered IV in Stage 2. Participants will receive the assigned dose of T-DXd until progression of disease or the participant meets one of the discontinuation criteria.

ELIGIBILITY:
KEY Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for randomization/registration into the study:

1. Adults aged ≥20 years in Japan, Taiwan, and Korea, or those aged ≥18 years in other countries, at the time the Informed Consent Forms (ICFs) are signed.
2. Pathologically-documented, unresectable, recurrent, or metastatic colorectal adenocarcinoma. Participants must have v-raf murine sarcoma viral oncogene homologue B1 (BRAF) wild-type cancer and rat sarcoma viral oncogenes homologue (RAS) status identified in primary or metastatic site.
3. The following therapies should be included in prior lines of therapy:

   1. Fluoropyrimidine, oxaliplatin, and irinotecan, unless contraindicated
   2. Anti-epidermal growth factor receptor (EGFR) treatment, if RAS wild-type and if clinically indicated
   3. Anti-vascular endothelial growth factor (VEGF) treatment, if clinically indicated
   4. Anti-programmed death ligand 1 (PD-(L)-1) therapy, if the tumor is microsatellite instability (MSI)-high/deficient mismatch repair (dMMR), or tumor mutational burden (TMB)-high, if clinically indicated
4. Confirmed human epidermal growth factor 2 (HER2)-overexpressing status assessed by central laboratory and defined as immunohistochemistry (IHC) 3+ or IHC 2+/ in situ hybridization (ISH) +.
5. Presence of at least one measurable lesion assessed by the Investigator per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
7. Has left ventricular ejection fraction (LVEF) ≥50% within 28 days before randomization/registration.

KEY Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Medical history of myocardial infarction (MI) within 6 months before randomization/registration, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV). Participants with troponin levels above the upper limit of normal (ULN) at Screening (as defined by the manufacturer), and without any MI-related symptoms, should have a cardiologic consultation before randomization/registration to rule out MI.
2. Has a corrected QT interval corrected with Fridericia's formula (QTcF) prolongation to >470 msec (female participants) or >450 msec (male participants) based on the average of the Screening triplicate 12-lead electrocardiograms (ECGs).
3. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
4. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within 3 months of the randomization/registration, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.).
5. Any autoimmune, connective tissue, or inflammatory disorders (eg, rheumatoid arthritis, Sjögren syndrome, sarcoidosis, etc.) where there is documented, or a suspicion of, pulmonary involvement at the time of Screening.
6. Prior pneumonectomy.
7. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole-brain radiotherapy and randomization/registration.
8. Participants with leptomeningeal carcinomatosis.
9. Has known human immunodeficiency virus (HIV) infection.
10. Active hepatitis B and/or hepatitis C infection, such as those with serologic evidence of viral infection within 28 days before study randomization/registration. Participants with past or resolved hepatitis B virus (HBV) infection are eligible if hepatitis B surface antigen (HBsAg) negative (-) and antibody to hepatitis B core antigen (anti-HBc) positive (+).

    Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
11. Previous treatment with a DXd-containing antibody-drug conjugate (ADC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (63):
- United States (9):
  - The University of Chicago, Chicago, Illinois
  - Norton Cancer Institute Audubon, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sarah Cannon (Tennessee Oncology - Nashville), Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Flinders Medical Centre (FMC), Bedford Park
  - Blacktown Hospital, Blacktown
  - Royal Brisbane & Women's Hospital, Brisbane
  - Monash Medical Centre, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
- Belgium (3):
  - UCL St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- France (8):
  - Hopital Jean Minjoz, Besançon
  - Hopital Edouard Herriot, Lyon
  - ICM-Val d'Aurelle, Montpellier
  - University Hospital of nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital St Antoine, Paris
  - Centre de Lutte Contre le Cancer CLCC - Institut Curie, Saint-Cloud
  - Chu Toulouse, Toulouse
- Italy (6):
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto Irccs, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Aienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda ULSS 8 Berica, Vicenza
- Japan (10):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kanagawa Cancer Center, Kanagawa
  - Kindai University Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- South Korea (6):
  - National Cancer Center (NCC), Goyang-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Clinico y Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall dHebron, Barcelona
  - Clinica Universitaria de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universitaria de Navarra, Pamplona
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital KMUH, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital CGMH - Kaohsiung Branch, Taoyuan District
  - Chang Gung Memorial Hospital-LinKou, Taoyuan District
- United Kingdom (5):
  - Beatson Glasgow, Glasgow
  - The Royal Marsden Hospital, London
  - UCLH Trust, London
  - The Christie, Manchester
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https:// vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: http://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Raghav K. Trastuzumab deruxtecan in HER2-positive advanced colorectal cancer: a plain language summary of the DESTINY-CRC02 study. Future Oncol. 2026 Jan;22(2):123-135. doi: 10.1080/14796694.2025.2606418. Epub 2026 Jan 5. PMID 41487064
- [Derived] Raghav K, Siena S, Takashima A, Kato T, Van den Eynde M, Pietrantonio F, Komatsu Y, Kawakami H, Peeters M, Andre T, Lonardi S, Yamaguchi K, Tie J, Castro CG, Hsu HC, Strickler JH, Kim TY, Cha Y, Barrios D, Yan Q, Kamio T, Kobayashi K, Boran A, Koga M, Allard JD, Yoshino T. Trastuzumab deruxtecan in patients with HER2-positive advanced colorectal cancer (DESTINY-CRC02): primary results from a multicentre, randomised, phase 2 trial. Lancet Oncol. 2024 Sep;25(9):1147-1162. doi: 10.1016/S1470-2045(24)00380-2. Epub 2024 Aug 5. PMID 39116902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 122 participants who met all inclusion criteria and no exclusion criteria were randomized/registered to T-DXd treatment in the United States, Asia-Pacific, and Europe.
Pre-assignment Details: Following adequate study explanation by the investigator or their designee, subjects voluntarily offered signed, informed consent prior to participation in any study procedures.
Groups:
- T-DXd 5.4 mg/kg Q3W: Participants were randomized to receive intravenous T-DXd administered at a dose of 5.4 mg/kg every 3 weeks (Q3W).
- T-DXd 6.4 mg/kg Q3W: Participants were randomized to receive intravenous T-DXd administered at a dose of 6.4 mg/kg every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Started | 82 | 40
Completed | 0 | 0
Not Completed | 82 | 40
Not completed — Adverse Event | 6 | 4
Not completed — Clinical Progression | 5 | 5
Not completed — Death | 2 | 1
Not completed — Other | 5 | 1
Not completed — Progressive Disease | 63 | 29
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W | Total
Number analyzed (Participants) | 82 | 40 | 122
Age, Categorical [Count of Participants; unit: Participants] — Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 54 | 23 | 77
    >=65 years | 28 | 17 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
  years | 58.5 (13.05) | 61.1 (12.13) | 59.3 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
  Participants
    Female | 37 | 21 | 58
    Male | 45 | 19 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
  Participants
    White | 35 | 15 | 50
    Black or African American | 0 | 0 | 0
    Asian | 42 | 24 | 66
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Blinded Independent Central Review Following IV Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2-overexpressing Metastatic Colorectal Cancer
Description: Confirmed objective response rate (ORR), defined as the number (percentage) of participants with complete response (CR) or partial response (PR), were assessed by blinded independent central review (BICR) based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as the disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: 6 months post-dose administration to data cut off, up to 20 months
Population: ORR was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
percentage of participants | 37.8 [27.3 to 49.2] | 27.5 [14.6 to 43.9]

2. Secondary Outcome: Confirmed Objective Response Rate by Investigator Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Overexpressing Metastatic Colorectal Cancer
Description: Confirmed objective response rate (ORR), defined as the number (percentage) of participants with complete response (CR) or partial response (PR), were assessed by Investigator assessment based on RECIST version 1.1. CR was defined as the disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. ORR was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From first dose administration to data cut off, up to approximately 19 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
percentage of participants | 31.7 [21.9 to 42.9] | 30.0 [16.6 to 46.5]

3. Secondary Outcome: Duration of Response Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Overexpressing Metastatic Colorectal Cancer
Description: DoR, defined as time from the initial response (CR or PR) by BICR and Investigator assessment until documented tumor progression or death from any cause. DoR was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From the first documented evidence of a response (complete or partial) until disease progression or death, up to approximately 19 months.
Population: DoR was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
months
  BICR | 5.5 [4.2 to 8.1] | 5.5 [3.7 to NA] — Not estimable due to insufficient data.
  Investigator | 5.6 [4.2 to 8.0] | 6.9 [4.9 to 9.9]

4. Secondary Outcome: Disease Control Rate Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2) -Overexpressing Metastatic Colorectal Cancer
Description: Disease Control Rate (DCR), defined as the proportion of subjects who achieved CR, PR, or SD for a minimum of 6 weeks during study treatment; DCR based on BICR and DCR based on Investigator assessments assessed according to RECIST version 1.1. DCR was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From first dose administration to data cut off, up to approximately 19 months.
Population: DCR was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
percentage of participants
  BICR | 86.6 [77.3 to 93.1] | 85.0 [70.2 to 94.3]
  Investigator | 89.0 [80.2 to 94.9] | 85.0 [70.2 to 94.3]

5. Secondary Outcome: Clinical Benefit Rate Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2) -Overexpressing Metastatic Colorectal Cancer
Description: Clinical Benefit Rate (CBR), defined as proportion of subjects who achieved CR, PR, or SD for at least 6 months; CBR based on BICR and CBR based on Investigator assessments will both be determined based on RECIST version 1.1. CBR was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From first dose administration to data cut off, up to approximately 19 months.
Population: CBR was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
percentage of participants
  BICR | 45.1 [34.1 to 56.5] | 32.5 [18.6 to 49.1]
  Investigator | 51.2 [39.9 to 62.4] | 42.5 [27.0 to 59.1]

6. Secondary Outcome: Progression Free Survival Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Overexpressing Metastatic Colorectal Cancer
Description: Progression Free Survival (PFS) defined as the time from date of randomization/registration until first objective radiographic tumor progression or death from any cause, based on BICR and Investigator assessment according to RECIST version 1.1. PFS was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From randomization to data cut off, up to approximately 19 months.
Population: PFS was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
month
  BICR | 5.8 [4.6 to 7.0] | 5.5 [4.2 to 7.0]
  Investigator | 5.8 [4.7 to 7.0] | 5.7 [4.2 to 8.3]

7. Secondary Outcome: Overall Survival Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Overexpressing Metastatic Colorectal Cancer
Description: Overall Survival (OS) defined as the time from date of randomization/ registration until death from any cause, according to RECIST version 1.1. OS was assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From randomization to data cut off, up to approximately 19 months.
Population: OS was assessed in the Full Analysis Set, which included 1 participant who was randomized/registered to T-DXd 6.4 mg/kg Q3W but actually received T-DXd 5.4 mg/kg Q3W.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 40
months | 13.4 [13.4 to 16.8] | NA [NA to NA] — Not estimable due to insufficient data.

8. Secondary Outcome: Percentage of Participants Reporting Treatment-emergent Adverse Events Following Intravenous Administration of T-DXd in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Overexpressing Metastatic Colorectal Cancer
Description: A Treatment-emergent Adverse Events (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug or has worsened in severity or seriousness after initiating the study drug until 47 days after the last dose of the study drug. Serious AEs with an onset or worsening 48 days or more after the last dose of study drug, if considered related to study treatment. are also TEAEs. TEAEs were assessed in the Safety Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From first dose administration to data cut off, up to approximately 19 months.
Population: The Safety Analysis Set (SAS) included all randomized/registered subjects who received at least 1 dose of study treatment. Subjects were summarized according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 83 | 39
percentage of participants | 98.8 | 100

9. Other Pre Specified Outcome: Change From Baseline in Patient-Reported Outcomes (PROs) in European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30)
Description: Exploratory outcome, results not included in this submission. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status/QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items and no item occurs in more than 1 scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Patient questionnaires were assessed in the Full Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From baseline to data cut off, up to approximately 19 months.
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Change From Baseline in Patient-Reported Outcomes (PROs) in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Colorectal Cancer 29 (QLQ-CR29)
Description: Exploratory outcome, results not included in this submission. EORTC QLQ-CR29 is designed to be administered in addition to EORTC QLQ-C30. The EORTC QLQ-CR29 is a specific questionnaire for Colorectal Cancer. Scale from 0 to 100, A higher scale represents better function and a higher quality of life.
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Patient-Reported Outcomes (PROs) in the EuroQol Questionnaire (EQ) of 5 Dimensions (5D) on a Standardized 5- Level (5L) Descriptive Health Status Scale (EQ-5D-5L)
Description: Exploratory outcome, results not included in this submission. The EQ-5D-5L is self-administered and consists of 2 parts, the EQ-5D-5L descriptive system and the EQ-visual analogue scale. On each dimension, a score of 1 indicates no patient problems in that dimension, 2 indicates slight problems in that dimension, 3 indicates moderate problems in that dimension, 4 indicates severe problems in that dimension and 5 indicates extreme problems in that dimension.
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Patient-Reported Outcomes (PROs) in Patient's Global Impression of Treatment Tolerability (PGI-TT)
Description: Exploratory outcome, results not included in this submission. The PGI-TT item is included to assess how a patient perceives the overall tolerability of the study treatment over the past 7 days. This is a single-item questionnaire, and patients will rate the bother associated with any treatment-related symptoms using response options ranging from "Not at all" to "Very much".
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Patient-Reported Outcomes (PROs) in Patient Global Impression of Symptom Severity (PGIS)
Description: Exploratory outcome, results not included in this submission. The PGIS item is included to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days. This is a single-item questionnaire, and patients will choose the response that best describes the severity of their overall cancer symptoms with options ranging from "No Symptoms" to "Very Severe".
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Patient-Reported Outcomes (PROs) in Patient Global Impression of Symptom Severity (PGIC)
Description: Exploratory outcome, results not included in this submission. The PGIC item is included to assess how a patient perceives their overall change in health status since the start of study treatment. This is a single-item questionnaire, and patients will choose from response options ranging from "Much Better" to "Much Worse".
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Inpatient Healthcare Resource Utilization
Description: Exploratory outcome, results not included in this submission. The impact of treatment and disease on healthcare resource use (including inpatient admissions, intensive care unit admissions, and length of stay in hospital) will be captured/collected in this study on an event-driven basis.
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: Exploratory outcome, results not included in this submission
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Serum Concentration of T-DXd
Description: Descriptive statistics will be provided for serum concentration data of T-DXd, DXd, and total anti-HER2 antibody. Serum concentrations were assessed in the Pharmacokinetics Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: C1D1 (Before infusion (BI), end of infusion (EOI) and 5 hours after infusion), C1D8 (7 days after infusion), C1D15 (14 days after infusion), C2D1 (BI and EOI), C3D1 (BI and EOI), C4D1, (BI and EOI), C6D1 (BI and EOI)
Population: The PK Analysis Set included all subjects randomized/registered in Stage 1 and/or Stage 2 who received at least 1 dose of T-DXd and had measurable serum concentrations of T-DXd. Subjects were analyzed according to the treatment received
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/L
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 83 | 39
ug/L
  C1D1 - Before Infusion: number analyzed (Participants) | 80 | 39
  C1D1 - Before Infusion | NA (NA) — Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC", NC = NA | NA (NA) — Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC", NC = NA
  C1D1 - End of Infusion: number analyzed (Participants) | 80 | 38
  C1D1 - End of Infusion | 118452.77 (27.5) | 134613.79 (18.1)
  C1D1 - 5Hrs After Infusion: number analyzed (Participants) | 76 | 38
  C1D1 - 5Hrs After Infusion | 123433.28 (23.0) | 142399.71 (19.8)
  C1D8 - 7 Days After Infusion: number analyzed (Participants) | 75 | 37
  C1D8 - 7 Days After Infusion | 22261.67 (38.9) | 28142.80 (51.5)
  C1D15 - 14 Days After Infusion: number analyzed (Participants) | 74 | 35
  C1D15 - 14 Days After Infusion | 8092.08 (61.7) | 11396.97 (60.3)
  C2D1 - Before Infusion: number analyzed (Participants) | 78 | 35
  C2D1 - Before Infusion | 2827.01 (118.8) | 4420.63 (73.0)
  C2D1 - End of Infusion: number analyzed (Participants) | 78 | 36
  C2D1 - End of Infusion | 109777.43 (67.2) | 135637.46 (22.2)
  C3D1 - Before Infusion: number analyzed (Participants) | 75 | 31
  C3D1 - Before Infusion | 4823.41 (83.6) | 7543.17 (74.3)
  C3D1 - End of Infusion: number analyzed (Participants) | 75 | 31
  C3D1 - End of Infusion | 122218.96 (25.8) | 139264.52 (24.7)
  C4D1 - Before Infusion: number analyzed (Participants) | 68 | 30
  C4D1 - Before Infusion | 5846.34 (89.5) | 11013.81 (51.8)
  C4D1 - End of Infusion: number analyzed (Participants) | 67 | 30
  C4D1 - End of Infusion | 124240.37 (23.4) | 134129.68 (30.3)
  C6D1 - Before Infusion: number analyzed (Participants) | 59 | 23
  C6D1 - Before Infusion | 7507.28 (74.5) | 10793.89 (59.0)
  C6D1 - End of Infusion: number analyzed (Participants) | 3 | 3
  C6D1 - End of Infusion | 117769.64 (25.3) | 35753.88 (1079.6)

17. Secondary Outcome: Serum Concentration of Total Anti-Human Epidermal Growth Factor Receptor 2 (HER2) Antibody
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/L
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 83 | 39
ug/L
  C1D1 - Before Infusion: number analyzed (Participants) | 80 | 39
  C1D1 - Before Infusion | 5211.18 (388.5) | 11934.79 (2058.9)
  C1D1 - End of Infusion: number analyzed (Participants) | 80 | 38
  C1D1 - End of Infusion | 110871.93 (28.8) | 121423.37 (20.3)
  C1D1 - 5Hrs After Infusion: number analyzed (Participants) | 76 | 38
  C1D1 - 5Hrs After Infusion | 107339.74 (23.4) | 124274.05 (23.0)
  C1D8 - 7 Days After Infusion: number analyzed (Participants) | 75 | 37
  C1D8 - 7 Days After Infusion | 27646.77 (40.3) | 32741.77 (49.9)
  C1D15 - 14 Days After Infusion: number analyzed (Participants) | 74 | 35
  C1D15 - 14 Days After Infusion | 10920.88 (71.7) | 14293.10 (63.0)
  C2D1 - Before Infusion: number analyzed (Participants) | 78 | 35
  C2D1 - Before Infusion | 3723.58 (123.1) | 4841.90 (107.5)
  C2D1 - End of Infusion: number analyzed (Participants) | 78 | 36
  C2D1 - End of Infusion | 106755.21 (66.0) | 127427.43 (23.2)
  C3D1 - Before Infusion: number analyzed (Participants) | 75 | 31
  C3D1 - Before Infusion | 6286.00 (93.2) | 9100.39 (90.0)
  C3D1 - End of Infusion: number analyzed (Participants) | 75 | 31
  C3D1 - End of Infusion | 114763.30 (22.8) | 134111.33 (19.5)
  C4D1 - Before Infusion: number analyzed (Participants) | 68 | 30
  C4D1 - Before Infusion | 7388.01 (101.8) | 14007.95 (67.2)
  C4D1 - End of Infusion: number analyzed (Participants) | 67 | 30
  C4D1 - End of Infusion | 113711.08 (21.5) | 133956.61 (30.5)
  C6D1 - Before Infusion: number analyzed (Participants) | 59 | 23
  C6D1 - Before Infusion | 9033.08 (94.9) | 13535.33 (73.5)
  C6D1 - End of Infusion: number analyzed (Participants) | 3 | 3
  C6D1 - End of Infusion | 104328.76 (35.4) | 37091.52 (816.2)

18. Secondary Outcome: Serum Concentration of Active Metabolite MAAA-1181a
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 83 | 39
pg/mL
  C1D1 - Before Infusion: number analyzed (Participants) | 80 | 39
  C1D1 - Before Infusion | NA (NA) — NA - Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC", NC = NA | NA (NA) — NA - Concentrations below the lower limit of quantitation (BLQ) are set to zero for the calculation of descriptive statistics. If any concentration at a time point is BLQ, the geometric mean at that time point is not calculated and is presented as "NC", NC = NA
  C1D1 - End of Infusion: number analyzed (Participants) | 80 | 39
  C1D1 - End of Infusion | 4101.40 (56.6) | 4313.38 (45.3)
  C1D1 - 5Hrs After Infusion: number analyzed (Participants) | 78 | 38
  C1D1 - 5Hrs After Infusion | 12063.71 (52.8) | 15773.44 (39.0)
  C1D8 - 7 Days After Infusion: number analyzed (Participants) | 73 | 37
  C1D8 - 7 Days After Infusion | 1372.33 (75.8) | 1761.02 (67.1)
  C1D15 - 14 Days After Infusion: number analyzed (Participants) | 75 | 35
  C1D15 - 14 Days After Infusion | 475.30 (62.4) | 602.43 (54.1)
  C2D1 - Before Infusion: number analyzed (Participants) | 79 | 35
  C2D1 - Before Infusion | 209.06 (74.6) | 291.07 (55.4)
  C2D1 - End of Infusion: number analyzed (Participants) | 80 | 36
  C2D1 - End of Infusion | 1474.48 (71.2) | 1649.91 (65.8)
  C3D1 - Before Infusion: number analyzed (Participants) | 75 | 33
  C3D1 - Before Infusion | 279.56 (64.0) | 427.33 (89.5)
  C3D1 - End of Infusion: number analyzed (Participants) | 74 | 32
  C3D1 - End of Infusion | 1559.93 (52.6) | 1647.92 (53.1)
  C4D1 - Before Infusion: number analyzed (Participants) | 68 | 30
  C4D1 - Before Infusion | 284.38 (81.4) | 494.17 (61.2)
  C4D1 - End of Infusion: number analyzed (Participants) | 67 | 30
  C4D1 - End of Infusion | 1448.53 (48.5) | 1404.67 (54.1)
  C6D1 - Before Infusion: number analyzed (Participants) | 59 | 23
  C6D1 - Before Infusion | 332.07 (81.3) | 578.72 (55.8)
  C6D1 - End of Infusion: number analyzed (Participants) | 3 | 2
  C6D1 - End of Infusion | 1182.53 (36.8) | 1512.25 (32.3)

19. Secondary Outcome: Percentage of Participants Positive for Treatment-emergent Anti-drug Antibodies (ADAs) and Neutralizing Antibodies (NAb) in Participants Who Were Administered T-DXd
Description: Immunogenicity will be assessed through characterization of incidence and titer of Anti-drug Antibodies (ADAs), the number and percentage of subjects positive for NAb of T-DXd by dose level will also be determined. ADAs and NAbs were assessed in the Immunogenicity Analysis Set at data cut-off date of 01 Nov 2022.
Time Frame: From baseline to data cut off, up to approximately 19 months
Population: The Immunogenicity Analysis Set included all subjects randomized/registered in Stage 1 and/or Stage 2 who received at least 1 dose of the study drug and who had at least
  1 baseline or postbaseline immunogenicity assessment. Subjects were analyzed according to the treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
Number analyzed (Participants) | 82 | 39
percentage of participants
  ADA | 1.3 | 0
  NAb | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug, up to approximately 44 months. For Final Results, data was collected up until 04 Dec 2024.
Description: Safety parameters were collected, analyzed, and reported based on the dosage of treatment drug administered as specified in the study protocol, therefore as 2 arms, T-DXd 5.4 mg/kg Q3W and T-DXd 6.4 mg/kg Q3W.
Arm/Group | T-DXd 5.4 mg/kg Q3W | T-DXd 6.4 mg/kg Q3W
All-Cause Mortality (participants affected / at risk) | 26/83 | 13/39
Serious Adverse Events (participants affected / at risk) | 21/83 | 12/39
Other Adverse Events (participants affected / at risk) | 81/83 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd 5.4 mg/kg Q3W (N=83) | T-DXd 6.4 mg/kg Q3W (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (4) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Inferior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd 5.4 mg/kg Q3W (N=83) | T-DXd 6.4 mg/kg Q3W (N=39)
Anaemia (Blood and lymphatic system disorders) | 22 (52) | 16 (43)
Neutropenia (Blood and lymphatic system disorders) | 8 (22) | 2 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 49 (102) | 22 (36)
Constipation (Gastrointestinal disorders) | 20 (20) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 19 (38) | 11 (14)
Vomiting (Gastrointestinal disorders) | 17 (29) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 12 (17) | 6 (13)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Asthenia (General disorders) | 17 (31) | 6 (20)
Fatigue (General disorders) | 16 (37) | 6 (9)
Pyrexia (General disorders) | 13 (19) | 4 (8)
Oedema peripheral (General disorders) | 5 (5) | 7 (8)
Malaise (General disorders) | 4 (5) | 5 (5)
Mucosal inflammation (General disorders) | 4 (4) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (4)
COVID-19 (Infections and infestations) | 14 (16) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 18 (39) | 16 (47)
Platelet count decreased (Investigations) | 18 (41) | 12 (25)
White blood cell count decreased (Investigations) | 11 (28) | 7 (22)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 7 (13)
Alanine aminotransferase increased (Investigations) | 8 (13) | 6 (12)
Blood creatinine increased (Investigations) | 4 (4) | 2 (3)
Lymphocyte count decreased (Investigations) | 4 (8) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 2 (4)
Blood bilirubin increased (Investigations) | 3 (5) | 6 (13)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 25 (41) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (8) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 8 (10) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dysgeusia (General disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (22) | 11 (12)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04744831/Prot_SAP_000.pdf